CLINICAL TRIAL: NCT03691792
Title: Optimizing Long-Term Outcomes for Winter Depression With CBT-SAD and Light Therapy: Confirming the Targets, Mechanisms, and Treatment Sequence
Brief Title: Optimizing Long-Term Outcomes for Winter Depression With CBT-SAD and Light Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: University of Pittsburgh (Other); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kelly Rohan, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH112819 (NIH)
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-06

CONDITIONS: Seasonal Affective Disorder
Keywords: cognitive-behavioral therapy; light therapy; biomarkers; treatment mechanisms
MeSH Terms: conditions — Seasonal Affective Disorder | interventions — Cognitive Behavioral Therapy; Phototherapy

STUDY DESIGN:
Intervention Model Description: head-to-head RCT
Who Masked: Outcomes Assessor
Masking Description: Outcomes are rated on a semi-structured interview by raters blind to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive-Behavioral Therapy (CBT-SAD) (Experimental): 12 1.5-hour group sessions at a rate of 2 sessions per week over 8 weeks.
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT-SAD)
- Light Therapy (Active Comparator): 6 weeks of daily light therapy at home, using a 10,000-lux light box beginning at 30 minutes upon waking, with dose subsequently adjusted per treatment algorithm.
  Interventions: Other: Light Therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy (CBT-SAD) — 12 group sessions over 6 weeks
  Other Names: CBT-SAD
  Arms: Cognitive-Behavioral Therapy (CBT-SAD)
Other: Light Therapy — 10,000-lux initiated at 30 min upon waking and adjusted per treatment algorithm, continuing for 6 weeks
  Arms: Light Therapy

SUMMARY:
Major depression is a highly prevalent, chronic, and debilitating mental health problem with significant social cost that poses a tremendous economic burden. Winter seasonal affective disorder (SAD) is a subtype of recurrent major depression that affects 5% of the population (14.5 million Americans), involving substantial depressive symptoms for about 5 months of each year during most years, beginning in young adulthood.

DETAILED DESCRIPTION:
Winter seasonal affective disorder (SAD) is a subtype of recurrent depression involving major depressive episodes during the fall and/or winter months that remit each spring. The central public health challenge in the management of SAD is prevention of winter depression recurrences. This application focuses on two SAD treatments that each work for some patients: light therapy (LT) and a SAD-tailored group cognitive-behavioral therapy (CBT-SAD). LT is the acute SAD treatment with the most substantial evidence to support its efficacy. Correction of circadian phase is LT's established target and mechanism. In our recently completed R01-level efficacy trial, post-treatment outcomes for CBT-SAD and LT were very similar, but CBT-SAD was associated with fewer depression recurrences over 2-year followup than LT (27.3% in CBT-SAD vs. 45.6% in LT). CBT-SAD engaged and altered a specific mechanism of action, seasonal beliefs, which improved at twice the rate during CBT-SAD compared to LT, and this improvement was associated with lower risk for recurrence following CBT-SAD. This confirmatory efficacy R01 will apply the experimental therapeutics approach to determine how each treatment works when it is effective and to identify the best candidates for each. We will ascertain whether theoretically-derived candidate biomarkers of each treatment's target and effect are prescriptive of better outcomes in that treatment vs. the other. Biomarkers of LT's target and effect include circadian phase angle difference (PAD) and the post-illumination pupil response (PIPR). Biomarkers of CBT-SAD's target and effect include pupil dilation and sustained gamma band EEG responses to seasonal words, which are hypothesized to reflect less engagement with seasonal stimuli following CBT-SAD and corroborate with the established target of seasonal beliefs. In addition to determining change mechanisms, we will test the efficacy of a "switch" decision rule upon recurrence to inform clinical decision-making in practice. We will randomize 160 adults with SAD to 6-weeks of CBT-SAD or LT in Winter 1; follow subjects in Winter 2; and, if a depression recurrence occurs, cross them over into the alternate treatment (i.e., switch from LT to CBT-SAD or CBT-SAD to LT). All subjects will be followed in Winter 3. Biomarker assessments will occur at pre-, mid-, and post-treatment in Winter 1, at Winter 2 followup (and again at mid-/post-treatment for those crossed-over), and at Winter 3 followup. Consistent with NIMH's priorities for demonstrating target engagement at the level of RDoC-relevant biomarkers, this work aims to confirm the targets and mechanisms of LT and CBT-SAD to maximize the impact of future dissemination efforts.

ELIGIBILITY:
Inclusion Criteria:

* Principle DSM-5 diagnosis of Major Depression, Recurrent, with Seasonal Pattern. -Meet Structured Interview Guide for the Hamilton Rating Scale for Depression-Seasonal Affective Disorder Version (SIGH-SAD) criteria for a current SAD episode (see below).
* No use or stable use of antidepressants (i.e., a consistent dose of the same medication maintained for > 4 weeks with no plans to change).

Exclusion Criteria:

* Current or past light therapy or CBT for SAD.
* Presence of a comorbid Axis I disorder that requires immediate treatment (i.e., bipolar disorder, psychotic disorders, substance use disorder).
* Acute and serious suicidal intent.
* Planned absences of >1 week from the area through March.
* History of conditions that are known contra-indications to LT, including conditions associated with toxicity of bright light to the retina (i.e., macular degeneration or any retinopathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Structured Interview Guide for the Hamilton Rating Scale for Depression-Seasonal Affective Disorder Version (SIGH-SAD) | past 1 week
  Semi-structured interview of depressive symptoms
Beck Depression Inventory-Second Edition (BDI-II) | past 2 weeks
  self-report measure of depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kelly J Rohan, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Psychology Department, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data will be provided to the NIMH Data Archive
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the study results.
URL: https://data-archive.nimh.nih.gov/

REFERENCES:
- [Derived] Rohan KJ, Franzen PL, Roeckelin KA, Siegle GJ, Kolko DJ, Postolache TT, Vacek PM. Elucidating treatment targets and mediators within a confirmatory efficacy trial: study protocol for a randomized controlled trial of cognitive-behavioral therapy vs. light therapy for winter depression. Trials. 2022 May 12;23(1):383. doi: 10.1186/s13063-022-06330-9. PMID 35550645